CLINICAL TRIAL: NCT05026398
Title: The Effect of Seven Day Fenfluramine Administration on Cognition in Healthy Volunteers
Brief Title: Fenfluramine and Cognition
Acronym: FEN&Cognition
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Zogenix International Limited, Inc., a subsidiary of Zogenix, Inc. (Industry); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Catherine Harmer, Prof Catherine Harmer, University of Oxford
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: FenCog
Record Dates: First submitted 2021-06-25; First posted 2021-08-30 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Cognitive Function
Keywords: Drug; Cognition; Dravet Syndrome; 5-HT; Sigma-1; Healthy Volunteers
MeSH Terms: conditions — Epilepsies, Myoclonic | interventions — Fenfluramine

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated to one of two groups (fenfluramine or placebo), stratified on group allocation, gender and cognitive task version administered. Participants in the fenfluramine group will receive oral solution of fenfluramine 15mg twice daily (BID) for seven days. Participants in the placebo group will receive a placebo oral solution 15mg twice daily (BID) for seven days. The study is assessing the effects of fenfluramine on cognitive ability, it is not an efficacy or safety study.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participant, Data Collectors, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Fenfluramine (Experimental): Drug: Fenfluramine - 15mg twice daily oral solution for seven days
  Interventions: Drug: Fenfluramine
- Placebo (Placebo Comparator): Placebo - 15mg twice daily oral solution for seven days
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Fenfluramine — Fenfluramine (30mg daily) will be dispensed in a cherry flavoured aqueous solution. Fenfluramine is both a serotonin releasing agent and sigma-1 receptor agonist. Fenfluramine is FDA approved for the treatment of Dravet syndrome, a rare form of epilepsy.
  Other Names: Fintepla (trade name); Fenfluramine Hydrochloride (ZX008)
  Arms: Fenfluramine
Other: Placebo — The placebo is a liquid designed to be identical to the interventional drug fenfluramine in terms of both taste and visual appearance. It will be administered at 30mg daily and dispensed in a cherry flavoured aqueous solution
  Arms: Placebo

SUMMARY:
In this study, the investigators will investigate the cognitive effects of fenfluramine, a drug that directly stimulates the release of serotonin in the brain and positively modulates σ1 function. The investigators will use fenfluramine to assess the cognitive effects of modulating serotonin and σ1 function in healthy volunteers using a battery of cognitive tasks that measure learning and memory, executive functioning, reward processing, and emotional processing. The study design is double-blind, and participants will be randomised to either seven days of fenfluramine or placebo administration. All participants will attend two screening visits to assess eligibility. There are two main study visits; during the first, participants will undertake cognitive tasks and questionnaires before taking the initial study dose. One the second study visit, participants will once again complete these tasks and questionnaires after a week of fenfluramine/placebo administration.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the research
* Not currently taking any medications (except the contraceptive pill)
* Aged 18-22 years
* Male or female
* Sufficiently fluent English to understand and complete the task
* Body Mass Index above 18-30
* Weight of 40-75kg

Exclusion Criteria:

* Current pregnancy (as determined by urine pregnancy test taken during Screening and First Dose Visit) or breast feeding
* Any past or current Axis 1 DSM-V psychiatric disorder
* Clinically significant abnormal values for liver function tests, clinical chemistry, urine drug screen, blood pressure measurement and ECG. A participant with a clinical abnormality or parameters outside the reference range for the population being studied may be included only if the Investigator considers that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures
* History of, or current medical conditions which, in the opinion of the investigator, may interfere with the safety of the participant or the scientific integrity of the study, including epilepsy/seizures, brain injury, hepatic or renal disease, severe gastro-intestinal problems, Central Nervous System (CNS) tumours, neurological conditions
* Current or past history of drug or alcohol dependency
* Current or past use of 3,4-Methylenedioxymethamphetamine (MDMA)
* Use of recreational drugs (e.g. cannabis, cocaine, amphetamines) within past 3 months
* Participation in a study which uses the same computer tasks as those in the present study (determined by asking participants about previous studies participated in during screening)
* Participation in a study that involves the use of a medication within the last three months
* Smoking > 5 cigarettes per day
* Typically drinks > 6 caffeinated drinks per day (e.g. tea, coffee, coca cola, Red Bull)
* Participant is unlikely to comply with the clinical study protocol or is unsuitable for any other reason, in the opinion of the Investigator

Ages: 18 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2022-06-22 (Actual)

PRIMARY OUTCOMES:
Change in Go/No-Go Task performance | Immediately before initial dose (Day 1) and immediately before final visit (Day 7)
  Accuracy on the Go/No-Go task
Change in Auditory Verbal Learning Task | Immediately before initial dose (Day 1) and immediately before final visit (Day 7)
  Accuracy on AVLT (number of items recalled across blocks)
Change in N-back task performance | Immediately before initial dose (Day 1) and immediately before final visit (Day 7)
  Accuracy on the N-back task

SECONDARY OUTCOMES:
Changes in reward sensitivity | Immediately before initial dose (Day 1) and immediately before final visit (Day 7)
  Sensitivity to reward as measured by the Probabilistic Instrumental Learning Task (PILT)
Changes in categorisation of emotional words | Immediately before initial dose (Day 1) and immediately before final visit (Day 7)
  Accuracy to categorise positive and negative descriptor words
Changes in recall of emotional words | Immediately before initial dose (Day 1) and immediately before final visit (Day 7)
  Number of words accurately recalled
Changes in recognition of emotional words | Immediately before initial dose (Day 1) and immediately before final visit (Day 7)
  Number of words accurately recognised
Changes in recognition of emotional facial expressions | Immediately before initial dose (Day 1) and immediately before final visit (Day 7)
  Accuracy of emotion labels (e.g. disgusted face) assigned by participants to expressive faces which have appeared on a computer screen for a period of 500ms.
Changes in visual short term memory on the Oxford Memory Test (OMT) | Immediately before initial dose (Day 1) and immediately before final visit (Day 7)
  Accuracy on the Oxford Memory Task
Changes in visual search ability | Immediately before initial dose (Day 1) and immediately before final visit (Day 7)
  Accuracy during contextual cueing task (CCT)
Changes in control measures of subjective state | Immediately before initial dose (Day 1) and immediately before final visit (Day 7)
  Ratings on the Positive and Negative Affect Schedule

CONTACTS AND LOCATIONS:
Overall Officials: Catherine J Harmer, DPhil, Principal Investigator — University of Oxford
Locations (1):
- Department of Psychiatry, University of Oxford, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data which has been fully de-identified may be shared with other academic and commercial organisations in the future, including those outside of the UK and the EU. Participants will be informed of this and specific consent to this is obtained within the Informed Consent Form.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: A few months after all data has been completed (ETA Jan 2022), unblinding has occurred (ETA Feb 2022), and all data analyses has been completed (ETA June 2022).
Access Criteria: The data will be made publicly available. Access requests will not be required.
URL: https://osf.io/x3t62/

DOCUMENTS (1):
  • Informed Consent Form (2021-07-28): https://cdn.clinicaltrials.gov/large-docs/98/NCT05026398/ICF_000.pdf